CLINICAL TRIAL: NCT03438773
Title: Prospective Pilot Feasibility Study Comparing Envarsus Once-a-day to Tacrolimus Twice-a-day Immunosuppressive Regimen on Drug Bioavailability in Hispanic First Time Kidney Transplant Recipients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: California Institute of Renal Research (Other)
Collaborators: Balboa Institute of Transplantation (Unknown); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VLX001-17; v01 01-Sep-2017 (Other: California Institute of Renal Research)
Record Dates: First submitted 2017-12-01; First posted 2018-02-20 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Kidney Transplant; Complications; Kidney Transplant Failure and Rejection
Keywords: Hispanic; First time kidney recipients
MeSH Terms: conditions — Rejection, Psychology | interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: Patients randomized into the study group will be prescribed Envarsus, mycophenolate and prednisone as a regimen vs. standard therapy with twice a day tacrolimus, mycophenolate and prednisone.
  Patients randomized to the control group will be prescribed standard immunosuppression with tacrolimus twice a day, anti-proliferative twice a day, and prednisone once a day at doses that are standard at our institution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Envarsus (Other): Study group - Envarsus once daily in addition to standard of care.
  Interventions: Drug: Envarsus
- Tacrolimus (Other): Control group - Tacrolimus twice daily in addition to standard of care.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Envarsus — Patients randomized into the Envarsus group will be prescribed Envarsus, mycophenolate and prednisone once daily.
  Arms: Envarsus
Drug: Tacrolimus — Patients randomized to the Tacrolimus group will be prescribed Tacrolimus twice-daily with standard of care immunosuppression, anti-proliferative and prednisone once-daily.
  Arms: Tacrolimus

SUMMARY:
This investigator-initiated post-marketing study will evaluate the role of Hispanic ethnicity on drug dosing of Envarsus in first-time stable renal transplant recipients. Tacrolimus trough drug levels will be studied as a primary endpoint at 24 hours after drug dosing and at steady state (e.g., trough level at 3 months post conversion) and secondary compliance assessments will be done by pill counts at clinic visits. Secondary outcomes will be the safety of once a day dosing as well as assessment of graft rejection and graft failure. In addition, concentration/dose ratios will be analyzed. The results of this study will provide important information about dosing of once a day tacrolimus (Envarsus) in Hispanic kidney transplant patients, which represents the largest growing group of patients with End-Stage Renal Disease

DETAILED DESCRIPTION:
Adequate drug dosing is essential to prevent allograft rejection and subsequent allograft loss. Many studies have shown that serum levels of immunosuppressant medications can be strongly influenced by the patient's genetic profile. Genetics has been shown to influence tacrolimus drug dosing in both liver and kidney transplant recipients 1. Whether these genetic differences influence care in clinical practice though is not known. Several genetic influences have been identified in Hispanic patients, such as polymorphisms in Cytochrome genes 1 and Nuclear Factor-kappa B genes 2, that might influence tacrolimus dosing and blood levels. In a study of Hispanic children, significant correlations were found to suggest that ethnic differences resulted in the need for higher or more frequent tacrolimus doing in Hispanic children 3. According to the Centers for Disease Control, Hispanics are 1.5 times as likely as non-Hispanic whites to develop ESRD 4 and Hispanics are the largest minority with the fastest growth of ESRD in the United States 5. Therefore it is likely that the unanswered question of whether there are differences in bioavailability of Envarsus in Hispanic patients will become even more relevant over time. Strategies that target improved bioavailability have the opportunity to significantly improve outcomes for all recipients of kidney transplants. Specifically, vulnerable patient populations, such as Hispanic patients, need to be studied to better understand the potential for altered bioavailability of immunosuppressive medications based on inherited pharmacologic traits.

Providing patients a once-a-day option for their immunosuppressive medication dosing is predicted to improve adherence, but whether once daily Envarsus provides adequate drug levels in Hispanic patient groups is not known. This study will carefully evaluate drug levels as a primary endpoint in this investigator-initiated study. Additional secondary outcomes to be measured over the two years of the study will be allograft rejection and allograft loss. The hypothesis of this study is that kidney transplant recipients receiving once-a-day extended release tacrolimus (Envarsus) will have outcomes that are not inferior to those who received twice-a-day tacrolimus during the two-year study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female 18 years of age or older.
* The subject is a first time stable renal transplant patients, who have received their transplant at least 3 months before study entry.
* The subject is willing to commit to the study design.
* The subject is considered to have stable allograft function defined as no documented rejection episodes within one month of screening.
* The subject is not currently receiving treatment with other experimental therapies directed at their transplant.

Exclusion Criteria:

* The subject has undergone a prior organ or bone marrow transplant.
* The subject has taken any interacting/contraindicated drug determined by the Investigator within 30 days of administration of the protocol.
* Any study drug allergies and if there are high serum donor specific antibody levels (DSA) or a high panel reactive antibody level (PRA).
* Documented treatment of rejection within 30 days of onset of the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-07-11 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Tacrolimus drug levels | 2 years
  Tacrolimus trough drug levels will be studied as a primary endpoint at 24 hours after drug dosing and at steady state through local lab HPLC MS/MS assays.

CONTACTS AND LOCATIONS:
Overall Officials: Arman Faravardeh, MD, Principal Investigator — California Institute of Renal Research
Locations (1):
- California Institute of Renal Research, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided